CLINICAL TRIAL: NCT05038904
Title: Preventing Life-Threatening Allergic Reactions With Acalabrutinib, an FDA-Approved Bruton's Tyrosine Kinase Inhibitor
Brief Title: Preventing Anaphylaxis With Acalabrutinib
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00223615
Record Dates: First submitted 2021-08-26; First posted 2021-09-09 (Actual); Results first posted 2023-09-28 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Food Allergy; Food Allergy Peanut
Keywords: Anaphylaxis; Peanut allergy; Tree nut allergy; Hypersensitivity
MeSH Terms: conditions — Food Hypersensitivity; Peanut Hypersensitivity; Anaphylaxis; Nut Hypersensitivity; Hypersensitivity | interventions — acalabrutinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib (Experimental): Participants will be given acalabrutinib (four doses of 100 mg of acalabrutinib to be taken orally twice daily).
  Interventions: Drug: Acalabrutinib

INTERVENTIONS:
Drug: Acalabrutinib — 100 mg oral capsule
  Other Names: Calquence

SUMMARY:
Food allergy is a potentially life-threatening condition, and its prevalence continues to increase despite public health efforts. There are currently no known therapies that can reliably prevent food-induced anaphylaxis. This is an open-label study designed to determine the ability acalabrutinib to prevent signs and symptoms of anaphylaxis during an oral food challenge in food-allergic adults.

DETAILED DESCRIPTION:
Approximately 15 million people (including 8% of children) in the US have a food allergy and are at risk for life-threatening systemic reactions to foods. There is an unmet need for treatments capable of preventing such reactions. This is a phase II, single-center, open label trial involving the use of acalabrutinib (brand name Calquence®) to prevent food-induced anaphylaxis in adults with food allergy. Acalabrutinib is FDA-approved to treat certain medical conditions, but it is not approved to treat allergies.

Adult participants with a physician-diagnosed food allergy to peanut and/or tree nuts will be enrolled. These participants will undergo an oral food challenge to peanut or a tree nut under close physician supervision to determine participants' baseline reactivity. After a rest period, the participants will take 4 oral doses of acalabrutinib 100 mg, and then repeat the oral food challenge to see if acalabrutinib will reduce participants' reactivity to peanut or tree nuts.

ELIGIBILITY:
Inclusion Criteria:

* History of immunoglobulin E (IgE)-mediated food allergy to peanut or tree nut
* Positive skin prick test to the trigger food (either peanut or tree nut)
* Objective clinical reaction to the food allergen during baseline oral food challenge
* Women of child bearing potential must agree to two forms of highly effective contraception (hormonal, device, or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and for 7 days following completion of acalabrutinib therapy.
* Ability to understand and the willingness to sign a written informed consent
* Ability to clearly understand and speak English at an 8th grade reading level

Exclusion Criteria:

* Participants who have been on immunomodulatory therapies or oral corticosteroids within 1 month prior to enrollment
* Participants with symptoms consistent with food reactions other than type 1 hypersensitivity
* History of allergic reaction to acalabrutinib
* History of idiopathic urticaria, dermatographism, idiopathic or unexplained anaphylaxis, or anaphylaxis (to foods or otherwise) resulting in intubation, prolonged hypotension, or neurological sequelae- History of cardiovascular disease
* History of a bleeding disorder, or those currently taking blood thinners
* History of stroke
* History of gastrointestinal ulcer
* History of cancer (other than skin cancer)
* Positive HIV status or history of other immunodeficiency
* Active or latent Hepatitis B or C infection based on laboratory testing
* Currently pregnant or nursing
* Current use of proton pump inhibitors (Note: participants currently receiving proton pump inhibitors who switch to H2-receptor antagonists or other antacids are eligible for enrollment to this study).
* Active significant infection
* Major surgical procedure within 28 days of enrollment
* Uncontrolled autoimmune hemolytic anemia or idiopathic thrombocytopenic purpura
* Difficulty swallowing oral medication, or significant gastrointestinal disease that would limit absorption of oral medication
* Concurrent participation in another therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-12-08 (Actual); Study Completion 2022-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melanie C. Dispenza, MD, PhD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Suresh RV, Dunnam C, Vaidya D, Wood RA, Bochner BS, MacGlashan DW Jr, Dispenza MC. A phase II study of Bruton's tyrosine kinase inhibition for the prevention of anaphylaxis. J Clin Invest. 2023 Aug 15;133(16):e172335. doi: 10.1172/JCI172335. PMID 37384412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: All study visits occurred between December 2021 and October 2022. Patients were recruited from the Johns Hopkins University Allergy and Clinical Immunology outpatient clinic and through IRB-approved advertising on social media. Patients who responded to advertisements were initially screened by telephone to determine eligibility. If determined eligible, patients were remote consented prior to Visit 1 by teleconference in compliance with FDA 21 CFR Part 11.
Pre-assignment Details: In this open-label trial, all eligible participants were given study drug.
Groups:
- Acalabrutinib: All participants received four oral doses of 100 mg of acalabrutinib twice daily.
Period: Overall Study
Arm/Group | Acalabrutinib
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 10
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 28 [23 to 36]
Sex/Gender, Customized [Count of Participants; unit: Participants] — Patients were asked to self-report their gender identity (options included male, female, and unspecified/ prefer not to answer).
  Participants
    Gender: Male | 5
    Gender: Female | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 9
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 10
Serum peanut-specific IgE [Median (Full Range); unit: kUA/L] | 4.9 [0 to 335]

OUTCOME MEASURES:

1. Primary Outcome: Highest Dose of Peanut That is Tolerated During Oral Food Challenge
Description: The highest dose of peanut protein (in mg) tolerated during oral food challenge before and after acalabrutinib treatment was determined by assessing clinical symptoms and physcial exam findings in each organ system during the challenge. Symptoms were given a numeric score based on the American Academy of Allergy, Asthma, and Immunology/European Academy of Allergy and Clinical Immunology PRACTALL consensus system to grade symptom severity and the likelihood of their representing a true objective clinical reaction to peanut.
Time Frame: Baseline and Day 2 of treatment
Measure: Median (Full Range); unit: mg
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 10
mg
  Baseline | 29 [1 to 444]
  Aftet treatment | 4,044 [444 to 4,044]
Statistical Analysis 1: Comparison: Acalabrutinib; Test type: Superiority — We estimated that 10 subjects allowed for 80% power to detect a 3-fold increase (1.1 natural log units; i.e. 1 food dose escalation) in the threshold food dose using a paired t test with p<0.05. For this sample size determination, the primary endpoint was assumed to be normally distributed with a standard deviation of 1.1 natural log units; p = 0.002, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Area Under the Curve Severity of Clinical Reaction to Peanut
Description: The severity of participants' cliinical reaction during oral food challenge before and after acalabrutinib treatment was determined using the American Academy of Allergy, Asthma, and Immunology/European Academy of Allergy and Clinical Immunology PRACTALL consensus system to grade objective clinical findings on physical exam on a scale of 0 (absent) to 3 (severe) in 9 different organ system categories. Total symptom scores for each food dose ranged from a minimum if 0 (no symptoms) to 27 (severe objective symptoms in all organ systems), and the area under the curve for all scores during the food challenge were calculated for each participant.
Time Frame: Baseline and Day 2 of treatment
Measure: Mean (95% Confidence Interval); unit: score on a scale*mg
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 10
score on a scale*mg
  Baseline | 27.83 [15.91 to 39.75]
  After treatment | 3.76 [0.12 to 7.39]
Statistical Analysis 1: Comparison: Acalabrutinib; Test type: Superiority; p = 0.0014, t-test, 2 sided

3. Secondary Outcome: Skin Prick Test Size to Peanut
Description: The skin prick test to peanut extract wheal area (in square mm) was measured at baseline and after treatment.
Time Frame: Baseline and Day 2 of treatment
Measure: Median (Full Range); unit: square mm
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 10
square mm
  Baseline | 126 [27.5 to 480]
  After treatment | 57.7 [0 to 345]
Statistical Analysis 1: Comparison: Acalabrutinib; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Basophil Activation Testing
Description: The percent of peripheral blood basophils activated by stimulation ex vivo with peanut extract was assessed by CD63 surface expression.
Time Frame: Baseline and Day 2 of treatment
Measure: Mean (Full Range); unit: percent of basophils activated
Arm/Group | Acalabrutinib
Number analyzed (Participants) | 10
percent of basophils activated
  Baseline | 31.7 [3.5 to 70.7]
  After treatment | 1.56 [0 to 4.6]
Statistical Analysis 1: Comparison: Acalabrutinib; Participants' ex vivo basophil activation during acalabrutinib treatment was compared to their own baseline level; Test type: Superiority; p = 0.002, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Description: This study followed the FDA Guidance For Industry ("Toxicity grading scale for healthy adult and adolescent volunteers enrolled in preventative vaccine clinical trials") grading system for adverse events.
Groups:
- Acalabrutinib: All participants who received acalabrutinib
Arm/Group | Acalabrutinib
All-Cause Mortality (participants affected / at risk) | 0/10
Serious Adverse Events (participants affected / at risk) | 3/10
Other Adverse Events (participants affected / at risk) | 5/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=10)
Sports-related concussion (Injury, poisoning and procedural complications) | 2 (2)
Sports-related injury (Injury, poisoning and procedural complications) | 1 (1)
Emergency room visit after baseline food challenge (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acalabrutinib (N=10)
Neutropenia (Blood and lymphatic system disorders) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 2 (2)
Elevated liver function tests (Hepatobiliary disorders) | 1 (1)
Eosinophilia (Blood and lymphatic system disorders) | 1 (1)
COVID-19 infection (Infections and infestations) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Hypokalemia (General disorders) | 1 (1)
Hypoalbuminemia (General disorders) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 2 (2)

LIMITATIONS AND CAVEATS:
Limitations included a small patient population, the lack of fully blinded oral food challenges, and the lack of placebo treatment arm. Additionally, this trial did not investigate alternative durations or dosages of acalabrutinib; therefore, the minimum effective duration and dose are as yet undetermined.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-09): https://cdn.clinicaltrials.gov/large-docs/04/NCT05038904/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-21): https://cdn.clinicaltrials.gov/large-docs/04/NCT05038904/ICF_001.pdf